CLINICAL TRIAL: NCT04935463
Title: Mucormycosis in COVID-19
Acronym: MUNCO
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Medanta Institute Delhi (Unknown); AIIMS Patna (Unknown); HCG Oncology Bangalore (Unknown); NSCB Jabalpur (Unknown)
Responsible Party: Principal Investigator, Shitij Arora, Associate Professor, Montefiore Medical Center
Other Study IDs: 2021-13086
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Covid19; Mucormycosis; Aspergillosis; Candida Infection
MeSH Terms: conditions — COVID-19; Mucormycosis; Aspergillosis; Candidiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose is to allow phsyician reporters to contribute to MUNCO registry. Mucormycosis in COVID-19 is a rapidly escalating medical emergency reported in high numbers in India during the ongoing coronavirus surge. There is very little known about the risk factors, patterns and complications of mucormycosis as it occurs either during the infection or treatment phase of the novel coronavirus (COVID-19). In light of this emerging epidemic within a pandemic, it is of time sensitive importance to obtain a better understanding of the risk factors and outcomes of this fatal complication

ELIGIBILITY:
Inclusion Criteria:

Diagnosed case of Mycotic Infection in COVID-19

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators have a web-based platform to allow physicians or other healthcare providers to report cases of confirmed Mucormycosis in patients with COVID 19. Physician reporters will individually enter de-identified data into a secure, electronic database (REDCap). The case report form will include items requesting the following information: age, country of residence, state of residence(within India), name of center/practice/physician reporting the case, gender, height, weight, patient's history specifics (diabetes, cancer, organ transplant, neutropenia, prior steroid use and intravenous drug use), COVID severity ( mild/moderate/severe), admission CRP values in mg/dL, COVID treatments prescribed, Mucormycosis treatment prescribed and site of mucormycosis( rhinocerebral, pulmonary, cutaneous or gastrointestinal) Once a reporter completes a survey, the reporter will not be able to access the survey again or update it
Sampling Method: Non-Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Vision loss | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided